CLINICAL TRIAL: NCT02218333
Title: Effect of Milk Proteins on Body Composition, Muscle Strength, Inflammation and Bone Health in Elderly Subjects
Brief Title: Health Effects of Milk Proteins in Elderly Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: The Research Council of Norway (Other); Tine (Industry); Oslo Metropolitan University (Other); Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Kirsten Holven, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014/150/REK sør-øst C
Record Dates: First submitted 2014-08-11; First posted 2014-08-18 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
MeSH Terms: interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control drink (Placebo Comparator): An isocaloric drink to milk
  Interventions: Dietary Supplement: Placebo
- Milk (Experimental): Protein enriched milk (Styrk)
  Interventions: Dietary Supplement: Milk

INTERVENTIONS:
Dietary Supplement: Milk — 4 dl milk will be consumed daily with breakfast and supper for 12 weeks
  Other Names: TINE Styrk milk
  Arms: Milk
Dietary Supplement: Placebo
  Other Names: Isocaloric drink
  Arms: Control drink

SUMMARY:
The aim of the present study is to investigate effects of milk on body composition and muscle strength, inflammation, appetite, DNA damage/repair and PBMC whole genome transcriptomics in elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 70 years of age
* reduced gait speed or
* reduced "five times sit to stand test" or
* reduced "timed step stair test " or
* reduced grip strength
* Stable body weight (last 3 months)
* Mini Nutritional Assessment (MNA®) score ≥ 17
* Mini-mental status (MMSE-NR) score: ≥ 24
* Willing to participate according to the protocol

Exclusion Criteria:

* Allergy/intolerance to milk/dairy products
* High intake of milk and yoghurt
* Physical active subjects
* Known diabetes type I or II, or HbA1c ≥ 6,5%
* Recent events of acute cardiovascular disease including stroke
* Rapidly evolving diseases (active malignancy) or history of cancer (malignant tumors) last 3 years.
* Severe inflammation-related diseases such as e.g. Crohn disease and arthritis
* Chronic obstructive pulmonary disease
* Increased blood pressure
* High intake of alcohol
* Reduced kidney function (GFR < 45 ml/min)
* Increased hsCRP, ASAT, ALAT
* Increased or suppressed TSH
* Hormone therapy
* Systemic use of glucocorticosteroids (anti-inflammatory steroid hormones). Use of spray and inhalator use is not exclusion.
* Disability preventing physical tests
* Using medications known to affect protein metabolism

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in muscle mass, strength and performance | Measured at baseline and after 12 weeks (end-of-study visit)
  Change in muscle is mass measured by DXA. Muscle strength and performance are measured by several physical tests such as repeated chair stands, handgrip strength, step stair test and strength in legs and torso and gait speed and are considered as the clinical relevant outcomes.

SECONDARY OUTCOMES:
Changes in levels of inflammatory markers | Measured at baseline and after 12 weeks (end-of-study visit)
  Changes in levels of inflammatory markers in circulation and at PBMC gene Expression Level such as i.e. CRP, IL-6, TNFa, IL-8, IL-18, ICAM, VCAM.

OTHER OUTCOMES:
Effect on PBMC whole genome transcriptomics | Measured at baseline and after 12 weeks (end-of-study visit)
  Measurement of PBMC Whole genome transcriptomics will be performed.
Changes in body composition (including bone mineral density) | Measured at baseline and after 12 weeks (end-of-study visit)
  Changes in body composition are measured by DXA.
Changes in the level of appetite regulatory hormones | Measured at baseline and after 12 weeks (end-of-study visit)
  Changes in the level of appetite regulatory hormones such as i.e. adiponectin, glucagon-like protein (GLP-1), gastric inhibitory polypeptide (GIP), ghrelin, Peptide YY (PYY) and cholecystokinin (CCK)
Changes in the Lymphocyte DNA damage and repair system | Measured at baseline and after 12 weeks (end-of-study visit)
  Changes will be measured using Whole blood and PBMC.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Holven, Professor, Principal Investigator — Institute of Basic Medical Sciences, Faculty of medicine, University of Oslo
Locations (1):
- University of Oslo, Oslo, Post Box 1046, Blindern, Norway

REFERENCES:
- [Derived] Gjevestad GO, Holven KB, Rundblad A, Flatberg A, Myhrstad M, Karlsen K, Mutt SJ, Herzig KH, Ottestad I, Ulven SM. Increased protein intake affects pro-opiomelanocortin (POMC) processing, immune function and IGF signaling in peripheral blood mononuclear cells of home-dwelling old subjects using a genome-wide gene expression approach. Genes Nutr. 2019 Nov 28;14:32. doi: 10.1186/s12263-019-0654-6. eCollection 2019. PMID 31798754
- [Derived] Ottestad I, Lovstad AT, Gjevestad GO, Hamarsland H, Saltyte Benth J, Andersen LF, Bye A, Biong AS, Retterstol K, Iversen PO, Raastad T, Ulven SM, Holven KB. Intake of a Protein-Enriched Milk and Effects on Muscle Mass and Strength. A 12-Week Randomized Placebo Controlled Trial among Community-Dwelling Older Adults. J Nutr Health Aging. 2017;21(10):1160-1169. doi: 10.1007/s12603-016-0856-1. PMID 29188875